CLINICAL TRIAL: NCT02010502
Title: Effects of Two Forms of Beetroot Juice Supplementation on Exercise Performance in Cyclists
Brief Title: Beet Root Supplement Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: J2013:089
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2018-04

CONDITIONS: Trained or Competitive Cyclists
Keywords: Beet root; exercise performance; cyclists

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Concentrated Beet Root Juice (Active Comparator): 500ml per day for 6 days
  Interventions: Dietary Supplement: Beetroot juice
- Beet root powder (Active Comparator): 500ml per day for 6 days
  Interventions: Dietary Supplement: Beetroot powder
- Placebo juice (Placebo Comparator): Negligible nitrate
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Beetroot juice
  Arms: Concentrated Beet Root Juice
Dietary Supplement: Beetroot powder
  Arms: Beet root powder
Dietary Supplement: Placebo
  Arms: Placebo juice

SUMMARY:
To examine the effects of two forms of beetroot juice supplementation on exercise performance in trained cyclists.

ELIGIBILITY:
Inclusion Criteria:

* good physical health
* trained or competitive cyclist
* between 18-40 years of age

Exclusion Criteria:

- have used any anabolic or ergogenic supplementation in the last 1-3 months

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Time to completion | Baseline to week 8

SECONDARY OUTCOMES:
O2 consumption | Baseline to Week 8

CONTACTS AND LOCATIONS:
Locations (1):
- Richardson Centre for Functional Foods and Nutraceuticals, Winnipeg, Manitoba, Canada